CLINICAL TRIAL: NCT04659148
Title: Surgical and Oncological Outcomes in Patients With Ulcerative Colitis Associated Rectal Cancer: a Retrospective Study
Brief Title: Surgical and Oncological Outcomes in Patients With Ulcerative Colitis-associated Rectal Cancer
Acronym: UC-RectalK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2712-2020
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Ulcerative Colitis; Rectal Cancer
Keywords: Ulcerative Colitis; Rectal Cancer
MeSH Terms: conditions — Colitis, Ulcerative; Rectal Neoplasms | interventions — Proctocolectomy, Restorative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total proctocolectomy — Total proctocolectomy: surgical removal of the colon, rectum, and anus

SUMMARY:
This is a retrospective observational study to investigate the short-term surgical outcomes, and long-term oncological outcomes of patients diagnosed with Ulcerative colitis and rectal cancer.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD) is a risk factor for the development of colorectal cancer (CRC). Despite improved targeted screening and timely prophylactic resection, up to 15% of all IBD-related mortality can be attributed to CRC.

Previous reports suggest that IBD patients present with CRC at an earlier age and with more advanced disease than those with sporadic CRC. The literature is limited, however, with respect to colitis-associated rectal cancer (CARC), which has unique considerations such as surgical approach and the use of neoadjuvant therapy. Although total proctocolectomy is generally the procedure of choice for those with CARC, recent reports reported acceptable oncological outcomes after ileal pouch-anal anastomosis (IPAA) and ileorectal anastomosis (IRA).

The impact of the type of surgical procedure on the oncologic outcome in patients with CARC is not well defined.

The aim of this study is to investigate short-term surgical outcomes (postoperative complications at 30 days after surgery) and long-term oncological outcomes (disease-free survival) of CARC patients undergoing different surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Ulcerative Colitis;
* Patients diagnosed with rectal cancer (within 15 cm from the anal verge);
* Patients who underwent surgery for rectal cancer between January 2004 and January 2020;
* All type of surgery will be included;
* Surgery in elective and emergency settings.

Exclusion Criteria:

* Patients aged<18 years;
* Patients with a diagnosis of undetermined colitis;
* Insufficient follow-up data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients with a proven diagnosis of Ulcerative Colitis and rectal adenocarcinoma, who underwent intestinal resection for curative intent, in elective or emergent setting, in the period between January 2004 and January 2020.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Surgical outcome | 30 days after surgery
  30 days postoperative complications
Oncological outcome | 5 years after surgery
  Disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — Istituto Clinico Humanitas
Locations (2):
- Humanitas Research Hospital, Rozzano, MI, Italy
- St. Mark's Hospital, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No